CLINICAL TRIAL: NCT03767322
Title: Effect of Allopurinol or Febuxostat to Prevent Contrast Induced Acute Kidney Injury (CI-AKI)
Acronym: CI-AKI
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Collaborators: Salvador López Gil (Unknown); Armando Vázquez Rangel (Unknown)
Responsible Party: Principal Investigator, Magdalena Madero, Nephrology Department, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PT-18-081
Record Dates: First submitted 2018-10-14; First posted 2018-12-06 (Actual); Last update posted 2018-12-06 (Actual); Status verified 2018-10

CONDITIONS: Contrast-induced Nephropathy; Contrast-induced Acute Kidney Injury
Keywords: contrast induced acute kidney injury; contrast induced nephropathy; allopurinol; febuxostat
MeSH Terms: interventions — Allopurinol; Febuxostat

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Allopurinol group (Active Comparator): The intervention group will receive 300 mg of allopurinol 12 hours before and 12 hours after the coronary intervention.
  Interventions: Drug: Allopurinol
- Placebo group (Placebo Comparator): The placebo group will receive 300 mg of placebo 12 hours before and 12 hours after the coronary intervention.
  Interventions: Drug: Placebo
- Febuxostat group (Active Comparator): The intervention group will receive 80 mg of febuxostat 12 hours before and 12 hours after the coronary intervention
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Allopurinol — Eligible patients will receive allopurinol 300 mg before and after coronary intervention
  Other Names: Zyloprim
  Arms: Allopurinol group
Drug: Febuxostat — Eligible patients will receive febuxostat 80 mg before and after coronary intervention
  Other Names: Turazive
  Arms: Febuxostat group
Drug: Placebo — Eligible patients will receive before and after coronary intervention
  Arms: Placebo group

SUMMARY:
A randomized, placebo-controlled, double-blind clinical trial of effect of allopurinol or febuxostat to prevent contrast induced acute kidney injury (CI-AKI)

DETAILED DESCRIPTION:
Eligible patients (patients with glomerular filtration rate < 60 ml/min or high riks patients based on Mehran score) that will be undergoing cardiac catheterization/intervention randomly assigned to receive allopurinol 300 mg or febuxostat 80 mg 12 hours before and 12 after 1 exposure of radiocontrast and IV hydration (normal saline 1 ml/kg/hr 12 pre and post radiocontrast exposure) or placebo and hydration.

Exclusion criteria: patients under treatment with allopurinol or febuxostat in the previous seven days, known allergy to allopurinol or febuxostat, patients on renal replacement therapy

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older who are scheduled to coronary intervention
* Patients with Mehran score > 5 or modified Mehran score >2 even glomerular filtration rate > 60 ml/min (high risk patients)
* Glomerular Filtration Rate < 60 ml/min
* All the patients provided written informed consent for the procedures and the test drug

Exclusion Criteria:

* Patients with shorter hospital stay (<48 hours)
* Patients under treatment with allopurinol of febuxostat
* Patients on renal replacement therapy
* Known allergy to allopurinol or febuxostat

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 558 (Estimated)
Dates: Start 2018-12-05 (Estimated); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Prevention of contrast induced acute kidney injury | 48 hours
  Increase in serum creatinine by ≥ 0.3 mg/dl within 48 hours

SECONDARY OUTCOMES:
Renal replacement therapy requirement | 7 days
  Initiation of renal replacement therapy
Length of hospitalization | 3 days to 90 days
  Length of hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Madero, MD, Principal Investigator — Instituto Nacional de Cardiologia Ignacio Chavez
Locations (1):
- Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, México City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ghelich Khan Z, Talasaz AH, Pourhosseini H, Hosseini K, Alemzadeh Ansari MJ, Jalali A. Potential Role of Allopurinol in Preventing Contrast-Induced Nephropathy in Patients Undergoing Percutaneous Coronary Intervention: A Randomized Placebo-Controlled Trial. Clin Drug Investig. 2017 Sep;37(9):853-860. doi: 10.1007/s40261-017-0542-z. PMID 28608311
- [Background] Kumar A, Bhawani G, Kumari N, Murthy KS, Lalwani V, Raju ChN. Comparative study of renal protective effects of allopurinol and N-acetyl-cysteine on contrast induced nephropathy in patients undergoing cardiac catheterization. J Clin Diagn Res. 2014 Dec;8(12):HC03-7. doi: 10.7860/JCDR/2014/9638.5255. Epub 2014 Dec 5. PMID 25653965
- [Background] Mendi MA, Afsar B, Oksuz F, Turak O, Yayla C, Ozcan F, Johnson RJ, Kanbay M. Uric Acid is a Useful Tool to Predict Contrast-Induced Nephropathy. Angiology. 2017 Aug;68(7):627-632. doi: 10.1177/0003319716639187. Epub 2016 Mar 22. PMID 27006404
- [Background] Shibagaki Y, Ohno I, Hosoya T, Kimura K. Safety, efficacy and renal effect of febuxostat in patients with moderate-to-severe kidney dysfunction. Hypertens Res. 2014 Oct;37(10):919-25. doi: 10.1038/hr.2014.107. Epub 2014 Jun 19. PMID 24942770
- [Background] Fukui T, Maruyama M, Yamauchi K, Yoshitaka S, Yasuda T, Abe Y. Effects of Febuxostat on Oxidative Stress. Clin Ther. 2015 Jul 1;37(7):1396-401. doi: 10.1016/j.clinthera.2015.03.026. Epub 2015 Apr 23. PMID 25913922